CLINICAL TRIAL: NCT07060339
Title: The Effect of Pain Coping Methods Used in the Active Phase of Labour on Birth Outcomes
Brief Title: Effect of Nonpharmacological Methods on The Active Phase Of Labour
Acronym: EFPCMUAPLBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Tuğba YILMAZ ESENCAN, assistant professor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-2/27
Record Dates: First submitted 2025-05-28; First posted 2025-07-11 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-06

CONDITIONS: Labour Pains; Massage; Exercise
Keywords: Labour Pain; Active Phase; Pain Management Techniques; Birth Experience; Midwifery Care
MeSH Terms: conditions — Labor Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study sample was divided into four groups: Group 1 - Intervention Group - (midwife monitoring during labour, breathing exercises, exercise and massage), Group 2 - Intervention Group - (midwife monitoring during labour, breathing exercises, massage and hot shower), Group 3 intervention group (midwife monitoring during labour, breathing exercises, exercise, massage and hot shower) and 4. intervention group (midwife monitoring during labour and pharmacological interventions). Data were collected face-to-face with a single midwife.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1. Intervention Group 1 - Exercise Programme (Experimental): Participants in this group were provided with midwifery care, breathing exercises, massage and exercise programmes during the active phase of labour. This group was formed to monitor the effects of exercise on the labour process.
  Interventions: Behavioral: Exercise Programme
- 2. Intervention Group 2 - Hot Shower Programme (Experimental): Participants in this group received midwifery care, breathing exercises, massage, and hot shower applications during the active phase of labour. This arm was designed to evaluate the effects of hot showers on labour pain, duration, and comfort.
  Interventions: Behavioral: Hot Shower Programme
- 3. Intervention Group 3 - Combined Application (Exercise + Hot Shower) (Experimental): In this group, midwifery care, breathing exercises, massage, exercise, and hot shower applications were applied together during the active phase of labour. This arm was designed to examine the effects of combining multiple non-pharmacological methods.
  Interventions: Behavioral: Combined Application (Exercise + Hot Shower)
- 4. Intervention Group - Pharmacological Intervention (Experimental): This group was monitored during the birth process with only midwifery care and routine pharmacological interventions. It serves as the standard care group that did not receive non-pharmacological interventions for comparison with other groups.
  Interventions: Behavioral: Pharmacological Intervention

INTERVENTIONS:
Behavioral: Exercise Programme — Midwifery care, breathing exercises, massage and exercise applications were performed on pregnant women in this group during the active phase of labour. Following breathing exercises, massage was applied for 10 minutes using different techniques according to rest and contraction intervals. Pain levels were assessed using the VAS before and after massage. After the massage, the exercise session began; the pregnant woman was first walked along a 50-metre corridor, followed by squatting, squat, four-legged positions, wall stretching movements, and pelvic tilt, swaying, and leg stretching exercises using a Pilates ball. Pain levels were measured using the VAS before and after all exercise applications.
  Arms: 1. Intervention Group 1 - Exercise Programme
Behavioral: Hot Shower Programme — In addition to midwifery care, breathing exercises, massage, and hot showers were administered in this group. Massage was administered for 10 minutes after the breathing exercises, and pain levels were measured using the VAS before and after the massage. After the massage, considering the risk of the pregnant woman falling, she was seated on a stool in the shower, and warm water at a temperature of 36.5-37.8 °C was applied to the lower abdomen and sacrum region during contractions for 15 minutes. To prevent chills, the application was repeated at 10-minute intervals, and pain levels before and after were again assessed using the VAS.
  Arms: 2. Intervention Group 2 - Hot Shower Programme
Behavioral: Combined Application (Exercise + Hot Shower) — In addition to midwifery care, breathing exercises, massage, exercise and hot shower treatments were performed for this group. As in Groups 1 and 2, the application began with breathing exercises, followed by massage, exercise, and hot showers in sequence. Pain levels were assessed using the VAS before and after each application, and measurements were taken again during the massage. Ten-minute breaks were given between applications to allow the pregnant women to rest, and the applications were continued alternately.
  Arms: 3. Intervention Group 3 - Combined Application (Exercise + Hot Shower)
Behavioral: Pharmacological Intervention — In this study, the fourth group was evaluated as the intervention 4 group and was followed up in accordance with standard interventions frequently applied during the birth process. Pregnant women in this group received routine midwifery care, massage treatments to promote relaxation, and breathing exercises in accordance with hospital protocols. In addition, pharmacological pain management methods commonly used in the clinic were also applied in this group.
  Arms: 4. Intervention Group - Pharmacological Intervention

SUMMARY:
The aim of this clinical trial is to evaluate the effects of methods such as exercise and hot showers applied during the active phase of labour on labour pain, labour duration, mode of delivery, newborn health, and the labour experience. In addition, the safety of these methods in terms of maternal and infant health will also be observed.

The main questions it aims to answer are:

Do exercise and warm shower applications reduce labour pain?

Do these methods shorten the duration of labour?

Is there a relationship between exercise and warm shower applications and the mode of delivery (vaginal birth/caesarean section)?

Do these practices affect the newborn's APGAR score?

Do women who use these methods have a more positive birth experience?

Participants:

Women who have started labour, are between 38 and 42 weeks pregnant, are expecting a single baby, and are having their first birth.

Participants will be randomly assigned to one of four groups:

Exercise

Warm shower

Exercise + warm shower

Pharmacological intervention (control group)

What is expected of participants:

Participate in exercise, warm shower, breathing exercises, and massage applications (depending on the group they are in) throughout the labour process

Participate in monitoring and evaluations during clinical check-ups

Complete postpartum questionnaires and scales related to the birth experience

This clinical study is being conducted to scientifically evaluate the effectiveness of non-pharmacological methods used during childbirth and to improve the birth experience.

DETAILED DESCRIPTION:
In the study, data were collected face-to-face with a single midwife. The data used in the study were the Informed Consent Form; the Informative Information Form developed by the researchers in line with the literature Information Form , the Birth Monitoring Form used during childbirth, the Visual Analogue Scale - VAS, the Postpartum Assessment Form, and the Birth Experience Scale.

ELIGIBILITY:
Criteria for Inclusion in the Study:

* In labour,
* Nulliparous,
* Cervical dilation greater than 3 cm,
* Full-term pregnancy (between 38 and 42 weeks of gestation),
* Carrying a single live foetus. *Reason for selecting nulliparous women: Multiparous women were excluded to randomise birth memory and avoid influencing case outcomes, as previous birth experiences may influence pain perception and birth experience.

Exclusion Criteria for Participants:

* Multiparity,
* High-risk pregnancies were not included in the study sample.

Ages: 18 Days to 45 Days | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — The study was conducted on primiparous pregnant women.
Enrollment: 120 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Visual Comparison Scale (Vizual Analogue Scale -VAS) | VAS is used repeatedly during the 4-5 cm, 6-7 cm, 8-9 cm and full dilation stages of labour, before and after massage, exercise and hot shower applications, and during intervention when necessary.
  VAS was used before and after each intervention to assess the level of pain during the birth process. Repeated measurements were taken between applications to monitor changes in pain and measure the effectiveness of the interventions.
Birth Experience Scale (BES) | By assessing her overall satisfaction with the birth process, it measures how she felt about the birth process and her physical and emotional experiences. It was completed within 24 hours after birth.
  It consists of 22 items and has 4 sub-dimensions.

CONTACTS AND LOCATIONS:
Locations (1):
- Üsküdar Üniversitesi Sağlık Bilimleri Fakültesi, İstanbul, Ümraniye 34662, Istanbul, Ümraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The study will be published in Yöktez.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The work started in January 2023 and ended in May 2025.
Access Criteria: The study can be accessed by entering Yöktez and typing the name of the study or the names of the administrators.
URL: https://tez.yok.gov.tr/UlusalTezMerkezi/

REFERENCES:
- See also: Gong, M., Dong, H., Tang, Y., Huang, W., & Lu, F. (2020). Aromaterapinin kaygı üzerindeki etkileri: Randomize kontrollü denemelerin meta analizi. Duygusal Bozukluklar Dergisi, 274, 1028-1040. — https://doi.org/10.1016/j.jad.2020.05.118
- See also: Uysal, C., Boz, İ., & Salman, S. (2022). Doğum Eyleminin Aktif Fazında Yaşanan Bel Ağrısının Yönetiminde Steril Su Enjeksiyonunun Etkisi: Randomize, Plasebo Kontrollü Bir Çalışma. Dokuz Eylül Üniversitesi Hemşirelik Fakültesi Elektronik Dergisi, 15(2), 1 — https://doi.org/10.46483/deuhfed.978831
- Available data/document: Individual Participant Data Set: non-pharmacological methods — https://dergipark.org.tr/tr/pub/ausbid/issue/38415/445612 — https://dergipark.org.tr/tr/pub/ausbid/issue/38415/445612